CLINICAL TRIAL: NCT05399420
Title: Study of the Quantitative Evolution of Circulating Cell-free DNA of Renal Origin in Patients With Acute Renal Failure
Brief Title: Study of Kidney Circulating Cell-free DNA in Patients With Acute Kidney Failure
Acronym: ADNIRA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CGenetix (Industry)
Collaborators: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: IDRCB 2022-A01259-34
Record Dates: First submitted 2022-05-25; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Kidney Failure, Acute
MeSH Terms: conditions — Acute Kidney Injury | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma sample (1 additional blood tube) from patients with functional kidney deficiency or organic kidney injury
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- functional kidney failure patients: Patients admitted to the nephrology department with suspicion of functional acute renal failures
  Interventions: Diagnostic Test: Blood sampling
- Organic kidney injury patients: Patients admitted to the nephrology department with suspicion of organic acute renal failure (kidney injury)
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — One additional blood tube will be collected for each patient included in the study using PAXgene Blood ccfDNA Tubes

SUMMARY:
The amount of total circulating DNA has been shown to increase in patients with acute renal failure. Nevertheless, it is currently not currently possible to prove the renal origin of this circulating DNA. Recently, in healthy subjects, teams have shown that it is possible to identify its tissue origin of circulating DNA. CGenetix is a MedTech company which develops on an identical principle an in vitro diagnostic test capable of identifying and quantifying renal degradation during an acute trauma. The objective of this study is to evaluate the sensitivity of the proposed technology to detect circulating DNA of renal origin released into the general circulation in patients with acute organic and functional renal failure. Patients with functional or organic kidney deficiency will be included and the kidney biomarkers develop by CGenetix will be compared between these 2 groups of patients.

DETAILED DESCRIPTION:
When the patient arrives, a first stage of checking the inclusion/non-inclusion criteria will be respected. Patients who do not meet the eligibility criteria will not be sampled (pre-screening stage).

Patients meeting the eligibility criteria will be informed of the study by the investigator and a written information note will be given to them. If they do not object to their participation, an additional tube of blood for research purposes will be taken during a blood sample taken as soon as they are admitted as part of their usual treatment. They will also follow the standard care protocol according to the clinical recommendations of their attending physician. The objective of early sampling is to sensitize the test by assaying the marker as soon as possible after renal injury. In the event of a posteriori differential diagnosis (obstructive ARF or IRC), the patient will be excluded from the final analysis.

Patients passing the pre-screening and screening stages positively will be included in the final analysis.

90 patients should be included and divided into 2 groups:

* 65 patients with non-biopsied organic acute kidney injury of which 20 patients with biopsied organic acute kidney injury (test group)
* 25 patients with functional acute kidney failure (control group).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Admitted for suspicion of acute renal injury (organic) and/or with an indication for renal biopsy (PBR)
* Patients hospitalized with functional acute renal failure (negative control and inclusion limited to n = 30 maximum)

Exclusion Criteria:

* Patients < 18 years old
* Patients with cognitive and mental disorders making them unable to express their non-objection to participation in the study
* Patients with obstructive renal failure
* Patients with chronic renal failure
* Patients who expressed their refusal to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in nephrology service for symptome suggesting a functional or organic kidney failure.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-09-10 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
Quantification of circulating cell-free DNA of renal origin at baseline (at patient hospital admission in nephrology department) | Patient hospitalization time
  Higher amount of circulating cell-free DNA of renal origin at the time of diagnosis of acute renal failure in patients with organ-type acute renal failure

SECONDARY OUTCOMES:
Comparison of circulating-cell-free DNA of renal origin amounts and kidney biopsy results at baseline (at patient hospital admission in nephrology department) | Patient hospitalization time
  Higher amount of circulating cell-free DNA of renal origin for patient with confirmed kidney lesions observed by histological analysis (kidney puncture)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Caudwell, MD, Principal Investigator — Centre Hospitalier Sud Francilien

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloom RD, Bromberg JS, Poggio ED, Bunnapradist S, Langone AJ, Sood P, Matas AJ, Mehta S, Mannon RB, Sharfuddin A, Fischbach B, Narayanan M, Jordan SC, Cohen D, Weir MR, Hiller D, Prasad P, Woodward RN, Grskovic M, Sninsky JJ, Yee JP, Brennan DC; Circulating Donor-Derived Cell-Free DNA in Blood for Diagnosing Active Rejection in Kidney Transplant Recipients (DART) Study Investigators. Cell-Free DNA and Active Rejection in Kidney Allografts. J Am Soc Nephrol. 2017 Jul;28(7):2221-2232. doi: 10.1681/ASN.2016091034. Epub 2017 Mar 9. PMID 28280140
- [Background] Merkle J, Daka A, Deppe AC, Wahlers T, Paunel-Gorgulu A. High levels of cell-free DNA accurately predict late acute kidney injury in patients after cardiac surgery. PLoS One. 2019 Jun 18;14(6):e0218548. doi: 10.1371/journal.pone.0218548. eCollection 2019. PMID 31211810
- [Background] Oellerich M, Sherwood K, Keown P, Schutz E, Beck J, Stegbauer J, Rump LC, Walson PD. Liquid biopsies: donor-derived cell-free DNA for the detection of kidney allograft injury. Nat Rev Nephrol. 2021 Sep;17(9):591-603. doi: 10.1038/s41581-021-00428-0. Epub 2021 May 24. PMID 34031575